CLINICAL TRIAL: NCT03192241
Title: PUMP (Providing the Underprivileged With Manual Pumps): A Randomized Controlled Trial
Brief Title: PUMP (Providing the Underprivileged With Manual Pumps): An RCT
Acronym: PUMP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: Academic Pediatric Association (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 1051735; 20170959 (Other: UC Davis)
Record Dates: First submitted 2017-06-16; First posted 2017-06-20 (Actual); Last update posted 2019-04-03 (Actual); Status verified 2019-04

CONDITIONS: Breastfeeding, Exclusive
Keywords: reading
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Intervention Model Description: Enrollment will be of 60 mother-infant dyads.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pump (Experimental): Mothers provided with a manual breast pump
  Interventions: Other: Pump
- book (Active Comparator): Mothers provided with a children's book
  Interventions: Other: Book

INTERVENTIONS:
Other: Pump — Intervention is providing mothers with a manual breast pump and instructions for when it could be used.
  Arms: Pump
Other: Book — Active control intervention is providing mother's with a children's book and information about reading to baby.
  Arms: book

SUMMARY:
The primary objective of this study is to pilot an intervention of providing manual breast pumps at hospital discharge to low-income, first-time mothers and to generate initial estimates of the effect of this intervention on exclusive breastfeeding rates at 3 months (12 weeks). In this pilot study, we will compare receipt of a breast pump and brief instructions of its use to the active control of receipt of a children's book and brief instructions about reading with baby. As a secondary objective, we will investigate mothers' attitudes and opinions about the manual breast pump intervention with the goal of fine-tuning it to best fit mothers' needs before a larger, multi-center trial. To support our objectives, we will examine the following specific aims:

1. To test the intervention of providing low-income, first time mothers with a manual breast pump at hospital discharge on exclusive breastfeeding rates at 12 weeks.

   Hypothesis: Among low-income first-time mothers, receipt of a manual breast pump at hospital discharge will lead to improved exclusive breastfeeding rates at 12 weeks postpartum compared to receipt of a children's book.
2. To use qualitative methods to determine best practices associated with successful implementation of a breast pump intervention to improve breastfeeding rates among low-income, first-time mothers.
3. To test the effect of receiving a children's board book during the birth hospitalization on parents reading to the baby at 3 months (12 weeks).

ELIGIBILITY:
Inclusion Criteria:

* WIC-eligibility (income below 185% the federal poverty line)
* liveborn infant
* in the well newborn nursery
* 12-96 hours of age
* infant is breastfeeding

Exclusion Criteria:

* maternal age <18 years
* maternal incarceration
* mother does not speak or read in English
* infant is a twin or higher level multiple
* infant has cleft lip and palate or a known syndrome

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2017-05-17 (Actual); Primary Completion 2019-01-30 (Actual); Study Completion 2019-01-30 (Actual)

PRIMARY OUTCOMES:
Exclusive breastfeeding at 12 weeks | 12 weeks
  Infant has had no food or drink other than breast milk in the last 24 hours

SECONDARY OUTCOMES:
Exclusive breastfeeding through 12 weeks | 12 weeks
  Infant has had no food or drink other than breast milk in their lifetime as measured at 12 weeks
Reading to baby at 12 weeks | 12 weeks
  Did parent read to baby in the last 24 hours & in the last week

OTHER OUTCOMES:
Exclusive breastfeeding at 6 weeks | 6 weeks
  Infant has had no food or drink other than breast milk in the last 24 hours
Any breastfeeding at 12 weeks | 12 weeks
  Infant has taken in breast milk in the last 24 hours
Any breastfeeding at 6 weeks | 6 weeks
  Infant has taken in breast milk in the last 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Laura R Kair, MD, Principal Investigator — University of California, Davis
Locations (1):
- University of California Medical Center, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hoyt-Austin AE, Cheng JH, Moua H, Tancredi DJ, Chantry CJ, Kair LR. Providing Low-Income Women With a Manual Pump: A Pilot Study. Hosp Pediatr. 2023 Feb 1;13(2):115-124. doi: 10.1542/hpeds.2021-006380. PMID 36646639